CLINICAL TRIAL: NCT05005143
Title: Improved Procedural Workflow For Catheter Ablation Of Paroxysmal AF With High Density Mapping System And Advanced Technology: DELETE AF Study
Brief Title: Improved Procedural Workflow For Catheter Ablation Of Paroxysmal AF With High Density Mapping System And Advanced Technology
Acronym: DELETE AF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: PI_2021/41
Record Dates: First submitted 2021-08-05; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Cardiac Arrhythmias; Atrial Fibrillation
Keywords: Catheter ablation; Arrhythmias; Mapping system; Atrial fibrillation
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paroxysmal AF ablation: Patients with standard indications to paroxysmal AF ablation

SUMMARY:
DELETE AF is a prospective, multicenter, non-randomized post-market study. All patients will be treated according to the standard care followed by each center. The protocol requires enrollment of consecutive patients from each center, according to eligibility criteria. During the 12 months follow-up period, clinical atrial fibrillation recurrence, occurrence of all kind of atrial arrhythmias and of all Adverse Events in the study population will be collected.

The purpose of this study is to demonstrate a low rate of clinical atrial arrhythmias recurrence with an improved procedural workflow for catheter ablation of paroxysmal AF, using the most advanced point-by-point RF ablation technology in a multicenter setting. The primary objective of the study is the rate of success at the medium-long term follow-up after PVI in a population of consecutive patients undergoing paroxysmal AF ablation. The success of the ablation is defined in terms of percentage of patients free from any clinical atrial arrhythmia at a 12-month follow-up from the procedure.

DETAILED DESCRIPTION:
Catheter ablation has been shown to be better than antiarrhythmic drug therapy in preventing clinical recurrences of atrial fibrillation (AF) and has emerged as an important therapeutic option for treating symptomatic drug-refractory, paroxysmal AF, with a Class I level A recommendation in ESC and ACC/AHA guidelines.

Improvements in ablation technologies and techniques to safely create more durable lesions and could improve the risk- benefit profile of this procedure. Recent advances in RF catheter design include models with real-time monitoring of catheter-to-tissue contact force. Evidence suggests improved clinical success in paroxysmal AF ablation with stable catheter-tissue contact. In addition, advances in diagnostic catheter manufacturing techniques have improved tissue contact and reduced interelectrode distances, allowing multipoint recording with high spatial resolution and improved signal fidelity. These algorithmic improvements have improved the signal-to-noise ratio and automated the validation of cardiac signals. Novel insights from this revolutionary ultra-high density (UHD) mapping with rapid acquisition of thousands of activation points deepened physiological and pathophysiological understanding of cardiac electrophysiology and arrhythmogenesis. This includes the cardiac conduction system itself and more importantly, due to the number of affected patients, the healthy and diseased working myocardium. In that sense HDM-based targeted ablation, in conjunction with pacing manoeuvres can be helpful to avoid excessive ablation. Moreover, HDM has also been found to allow greater precision in the identification of reconnection gaps in pulmonary veins, therefore, targeted ablation resulted in lower radiofrequency time for PVI. The technological advances present great opportunities for improving the electroanatomic characterization of low-voltage activity in tissue such as the PV antra, likely representing vulnerabilities in antral lesion sets, and ablation of these targets seems to improve freedom from AF

The primary objective of the study is the rate of success at the medium-long term follow-up after PVI in consecutive patients undergoing atrial fibrillation ablation. The success of the ablation is defined in terms of percentage of patients free from any clinical atrial arrhythmia at a 12-month follow-up from the procedure.

Secondary objectives of the study are: evaluation of acute procedural success, correlation between acute success and medium- long-term success, evaluation of the proportion of patients who will be asymptomatic during follow-up, patient reported outcomes, rate of clinical atrial fibrillation recurrence during follow up, rate of occurrence of other arrhythmias during follow-up, association between occurrence of atrial arrhythmias and baseline patient's characteristics (clinical history and drug therapy) or procedural data (post-hoc voltage and activation maps analysis), estimation of costs associated with the use of health care resources, rate of the adverse events associated with the primary ablation procedure and overall procedure time.

ELIGIBILITY:
Inclusion Criteria:

* History of recurrent symptomatic paroxysmal AF (PAF) with ≥1 episode reported and documented within the 365 days prior to enrollment; PAF is defined as AF episodes that last ≥30 seconds in duration and terminate within 7 days.
* Patients with an indication to an ablation procedure with 3D high-density mapping system according to current international and local guidelines (and future revisions), existing IFU and per physician discretion
* Patients who are willing and capable of providing informed consent, participating in all testing at an approved clinical investigational center.
* Patients whose age is 18 years or above, and of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

* Patients who have persistent or long-standing persistent AF (>1 AF episodes lasting greater than 7 days, with no episodes having lasted greater than 30 days, within the past year)
* Patients who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments
* Patients who are unwilling or unable to sign an authorization to use and disclose health information or an Informed Consent.
* Patients unavailable or not willing to complete follow up visits and examination for the duration of the study at the center.
* Life expectancy ≤ 12 months per physician judgment.
* Patients who have undergone a previous cardiac ablation within 90 days prior to enrollment;
* Unrecovered/unresolved Adverse Events from any previous invasive procedure;
* Women of childbearing potential who are, or plan to become, pregnant during the time of the study (method of assessment upon physician's discretion)
* Left atrial size > 60 mm diameter on echocardiogram
* Left atrial thrombus in pre-procedure imaging within 4 weeks of the ablation procedure.
* AF secondary to electrolyte imbalance, thyroid disease or reversible non- cardiac cause.
* History of prior surgical ablation for AF or atypical atrial flutter, including MAZE or mini MAZE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients, clinically indicated for paroxysmal AF ablation, will be enrolled after signing an informed consent form and an authorization to use and disclose health information.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number and percentage of patients with clinical atrial arrhythmia recurrences | 12 months
  The primary outcome measure of this study is to estimate, after 12-months from the procedure, the number and the percentage of patients with documented clinical atrial arrhythmia recurrences. Arrhythmias in the definition are any AF, atrial flutter, or atrial tachycardia episode, continuous for >30 seconds, as recorded by any post-ablation ECG modality. Arrhythmia recurrences within the first 3 months (blanking period) are classified as early recurrences and will not be considered procedural failure

SECONDARY OUTCOMES:
Acute procedural success of AF ablation | Within 30 minutes after ablation procedure
  This secondary outcome measures the percentage of acute procedural success. The acute success of the AF ablation is verified by: the completion of the necessary ablation application(s), the validation of ablation through appropriate technique(s) and, when applicable, the termination of the primary arrhythmia.
Baseline patient's characteristic (clinical history and drug therapy) for subjects undergoing catheter ablation | 12 months
  This secondary outcome measures the baseline patient's characteristics (clinical history and drug therapy) as potential predictors of primary arrhythmia recurrences, that will be evaluated at 12 months
Procedural ablation parameters | Intraoperative
  This secondary outcome measures the radiofrequency delivery time, the total ablation time, the fluoroscopy time, acquisition time, number of points per map, cardiac area and volume acquired from the maps
Rate of adverse events and complications during procedure and follow up | 12 months for adverse events during follow up and intraoperative for acute adverse events
  This secondary outcome measures the rate of the adverse events that occurs during the procedure and after 12 months
Estimate costs related to the use of health care resources | 12 months
  This secondary outcome measures the resource consumption and the associated costs in term of ablation procedures, follow-up, management of complication and health care resources utilization
Patient reported outcomes: EQ-5D-5L | 12 months
  This secondary outcome measures patient reported outcomes through specific symptom scale questionnaire: EQ-5D-5L score will be obtained as the sum of units on the questionnaire's scale
Patient reported outcomes: EHRA Score of AF-related Symptoms | 12 months
  AF related symptoms and symptom burden will be measured through the Symptom Severity Questionnaire and EHRA Symptom Classification Score of AF-related Symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Garcia-Bolao, Principal Investigator — Department of Cardiology and Cardiac Surgery, Clínica Universidad de Navarra

REFERENCES:
- [Derived] Solimene F, Stabile G, Ramos P, Segreti L, Cauti FM, De Sanctis V, Maggio R, Ramos-Maqueda J, Mont L, Schillaci V, Malacrida M, Garcia-Bolao I. Improved procedural workflow for catheter ablation of paroxysmal AF with high-density mapping system and advanced technology: Rationale and study design of a multicenter international study. Clin Cardiol. 2022 Jun;45(6):597-604. doi: 10.1002/clc.23806. Epub 2022 Apr 21. PMID 35446440